CLINICAL TRIAL: NCT00512564
Title: Clinical and Laboratory Assessment of Iron Overload in Sickle Cell Anemia and Sickle Cell Thalassemia - An Observational and Laboratory Study
Brief Title: Clinical and Laboratory Assessment of Iron Overload in Sickle Cell Anemia and Sickle Cell Thalassemia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0087-07-EMC
Record Dates: First submitted 2007-08-05; First posted 2007-08-07 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Sickle Cell Anemia; Sickle Cell Thalassemia
Keywords: Sickle Cell Anemia; Sickle Cell Thalassemia; Iron overload; Non transferrin binding iron; Hepcidin
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients suffering from Sickle cell disease
  Interventions: Other: Laboratory analyses of iron overload

INTERVENTIONS:
Other: Laboratory analyses of iron overload — Summary of clinical status related to iron overload and laboratory analysis of Iron overload including Total serum Iron, Transferrin, Ferritin and Non transferrin Binding Iron and Labile Plasma Iron

SUMMARY:
Iron overload is well study in Thalassemia patients and it's not only related to blood transfusions, since intestinal iron absorption is also increased in those patients. Sickle cell patients didn't developed significant clinical symptoms and signs of iron overload in spite frequent transfusions. The purpose of this study is to assess the iron overload in Sickle cell anemia and Sickle cell Thalassemia patients using clinical parameters and laboratory studies including Non Transferrin Binding Iron, Labile Iron and Hepcidin, in order to determine the cardiac and liver iron.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with Sickle Cell Anemia and Sickle Cell Thalassemia that are treated and followed up at the Pediatric Hematology Unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All tha patinets suffering from Sickle cell disease trreated at the Pediatric Hematology Unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Hematology Unit, Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Afula, Israel